CLINICAL TRIAL: NCT05286619
Title: A Study of Pembrolizumab (MK-3475) Plus Platinum and Gemcitabine as First Line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (PIPER)
Acronym: PIPER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Cancer Research Malaysia (Other); Kuala Lumpur General Hospital (Other Government); National Cancer Institute, Malaysia (Other Government); Merck Sharp & Dohme LLC (Industry); My Starfish Foundation (Unknown); Yayasan Sime Darby (Unknown); Yayasan PETRONAS (Unknown)
Responsible Party: Principal Investigator, A/Prof. Dr. Wan Zamaniah Wan Ishak @ Wan Mohammad, Associate Professor Dr, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CRMY(HN)2021001
Record Dates: First submitted 2022-02-11; First posted 2022-03-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus Platinum and Gemcitabine (Experimental): Pembrolizumab 200 mg will be administered as 30-minute IV infusion Day 1 of every 3 weeks. Pembrolizumab will be administered first followed by the platinum and gemcitabine infusions. Cisplatin will be administered on Day 1 and 8 of each 3-weeks treatment cycle with a dose of 35 mg/m2 for 60 minutes. Carboplatin will be administered on Day 1 of each 3-weeks treatment cycle given as a dose of AUC 5 for 60 minutes. Gemcitabine will be administered on Day 1 and 8 of each 3-weeks treatment given as a dose of 1250 mg/m2 for 30 minutes. AEs associated with pembrolizumab exposure, including coadministration with additional compounds, may represent an immunologic aetiology. If one or all of the chemotherapy components is discontinued, subjects can continue with pembrolizumab up to the full 35 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg will be administered on Day 1 every 3 weeks for up to 24months
Drug: Cisplatin — Cisplatin at 35 mg/m2 IV using a split dose regimen on Day 1 and Day 8 of each 3-week cycle, up to 6 cycles.
Drug: Carboplatin — Carboplatin at AUC 5 IV on Day 1 of each 3-week cycle, up to 6 cycles.
Drug: Gemcitabine — Gemcitabine 1250mg/m2 IV on Day 1 and Day 8 of each 3-week cycle, up to 6 cycles

SUMMARY:
This is an open-label, single-arm, Phase 2 study of pembrolizumab plus platinum and gemcitabine (PG) in subjects with recurrent or metastatic head and neck cancer squamous cell carcinoma (R/M HNSCC). Evaluable 63 subjects with R/M HNSCC will be enrolled for examination of the efficacy and safety of the combination of pembrolizumab (200 mg IV on Day 1 of each 3-week cycle, up to 35 cycles) in combination with platinum (either cisplatin at 35 mg/m2 IV using a split-dose regimen on Day 1 and Day 8 or carboplatin at AUC 5 IV on Day 1 of each 3-week cycle, up to 6 cycles) and gemcitabine at 1250 mg/m2 IV on Day 1 and 8 of each 3-week cycle, for up to 6 cycles as first-line treatment. This study will be conducted in conformance with Good Clinical Practices. Specific procedures to be performed during the trial, as well as their prescribed timelines and associated visit windows, are outlined in the protocol.

DETAILED DESCRIPTION:
This is an open label, single arm, Phase 2 study of pembrolizumab plus platinum and gemcitabine (PG) in subjects with recurrent or metastatic head and neck cancer squamous cell carcinoma (R/M HNSCC) to be conducted in conformance with Good Clinical Practices. Evaluable 63 subjects with R/M HNSCC will be enrolled for examination of the efficacy and safety of the combination of pembrolizumab with PG as first line treatment.

The purpose of the study is to determine Pembrolizumab in combination with platinum and gemcitabine chemotherapies would be comparable with or better than the combination of pembrolizumab with platinum plus 5-FU chemotherapies, in terms of objective response rate(ORR), overall survival (OS) and safety as first-line treatment in R/M HNSCC.

All subjects will be given pembrolizumab (200 mg IV on Day 1 of each 3-week cycle, up to 35 cycles) in combination with platinum (either cisplatin at 35 mg/m2 IV using a split dose regimen on Day 1 and Day 8 or carboplatin at AUC 5 IV on Day 1 of each 3-week cycle, up to 6 cycles) and gemcitabine at 1250 mg/m2 IV on Day 1 and 8 of each 3-week cycle, for up to 6 cycles. Disease status will be followed by imaging studies at 6 weekly intervals (±7 days) during the first year, and every 9 weeks (±7 days) after the first year, until disease progression, withdrawal of consent, death or end of study. RECIST 1.1 will be used as the primary efficacy endpoint of response rate. Safety will be monitored according to the National Cancer Institute CTCAE Version 5.0.

Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the protocol under section Schedule of Activities (SoA).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of R/M HNSCC that is considered incurable by local therapies will be enrolled in this study:

   * Subject may not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy which was completed more than 6 months prior to signing consent if given as part of multimodal treatment for locally advanced disease is allowed.
   * The eligible primary tumour locations are oropharynx, oral cavity, hypopharynx, and larynx.
   * Subject may not have a primary tumour location site of nasopharynx (any histology).
2. A male participant must agree to use a contraception as detailed in Appendix 3: Contraceptive Guidance and Pregnancy Testing of this protocol starting with the first dose of study treatment through the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant (see Appendix 3: Contraceptive Guidance and Pregnancy Testing), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3: Contraceptive Guidance and Pregnancy Testing OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3: Contraceptive Guidance and Pregnancy Testingduring the treatment period and for at least 180 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) willing and able to provides written informed consent for the trial. The participant may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Archival or fresh tumor tissues must be available for evaluating relevant biomarkers. Newly obtained core needle or excisional biopsy of a tumor lesion not previously irradiated is preferred to archived tissue. If newly obtained samples cannot be obtained due to inaccessibility or patient safety concern, submission of paraffin block or formalin-fixed, paraffin embedded (FFPE) slides of up to 3 years prior to trial enrolment are acceptable (15 unstained slides of 5 microns in thickness). Refer to Section 6.1.5 for complete information on the tissue sample collection.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
8. Have adequate organ function as defined in the following table (Table 3). Specimens must be collected within 10 days prior to the start of study intervention.

   * Absolute neutrophil count (ANC) ≥1500/µL
   * Platelets ≥100 000/µL
   * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
   * Creatinine ≤1.5 × ULN
   * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
   * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
   * International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Has disease that is suitable for local therapy administered with curative intent.
2. Has progressive disease within six months of completion of curatively intended treatment for locoregionally advanced HNSCC.
3. Patient with an expected life expectancy of less than 3 months.
4. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment allocation (see Appendix 4). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
5. Has received prior therapy with an anti-PD-1, anti-PD-L1, or antiPDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137).
6. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to start of study treatment.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
7. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
8. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
12. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
15. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
16. Has an active infection requiring systemic therapy.
17. Has a known history of Human Immunodeficiency Virus (HIV) infection.
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
22. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  To determine Objective Response Rate (ORR) per RECIST 1.1 to treatment of pembrolizumab plus platinum and gemcitabine in recurrent/metastatic (R/M) head and neck squamous cell carcinoma (HNSCC) patients.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  1) To evaluate the Overall Survival (OS) to combination treatment of pembrolizumab plus platinum and gemcitabine in R/M HNSCC patients
Incidence of Treatment-Related Adverse Events (Safety and tolerability) | 24 months
  To evaluate the number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Progression Free Survival (PFS) | 24 months
  2) To estimate Progression Free Survival (PFS) per RECIST 1.1 to combination treatment of pembrolizumab plus platinum and gemcitabine in R/M HNSCC patients
Response duration (DOR) | 24 months
  3) To estimate response duration (DOR) per RECIST 1.1 to combination treatment of pembrolizumab plus platinum and gemcitabine in R/M HNSCC patients
ORR and OS correlation | 24 months
  To evaluate the ORR and OS in correlation with PD-L1 Combined Positive Score (CPS)

OTHER OUTCOMES:
Genetic variation | 24 months
  To explore correlation between genetic variation and clinical response of patients.
Microbiome profiling | 24 months
  To conduct on-treatment microbiome profiling and determine the correlation with clinical response
Circulatory immune cells correlations | 24 months
  To explore the changes in circulatory immune cells throughout the treatment period of patients

CONTACTS AND LOCATIONS:
Overall Officials: Wan Zamaniah Wan Ishak, MBBS, MD, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Manuscript specific data will be shared with qualified external researches, access to patient-level data. These requests can be made via email to principal investigator of the study. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable law and regulations.
Supporting Information: Study Protocol
Time Frame: From 22 Sept 2022 till June 2026
Access Criteria: Manuscript specific data will be shared with qualified external researches, access to patient-level data. These requests can be made via email to principal investigator of the study. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable law and regulations.

REFERENCES:
- [Derived] Cheong SC, Selvam B, Ho GF, Muhamad Nor I, Tan CK, Wong YF, Teo SH, Lim KP, Chai AWY, Yahya A, Wan Ishak WZ. Pembrolizumab (MK-3475) plus platinum and gemcitabine as first-line treatment of recurrent/metastatic head and neck squamous cell carcinoma (PIPER): a phase 2, multicentre, single-arm protocol study in Malaysia. BMJ Open. 2024 Dec 3;14(12):e076898. doi: 10.1136/bmjopen-2023-076898. PMID 39627139